CLINICAL TRIAL: NCT01231945
Title: Low-Cost Molecular Cervical Cancer Screening Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911015; 11-C-N015
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-12-20

CONDITIONS: DNA Probes; E6 Protein; Uterine Cervical Neoplasms; HPV
Keywords: Cervical Cancer; Human Papilloma Virus (HPV); Cervical Intraepithelial Neoplasia (CIN)
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Low-cost molecular human papillomavirus (HPV) testing may offer a more robust alternative to Pap smears and visual inspection for cervical cancer screening of underserved women. Two low-cost molecular tests for human HPV, the HPV E6 Test and the careHPV test, have been developed to detect cervical cancer by testing for HPV DNA. These tests take between 2 and 3 hours to run and may provide point-of-care (diagnostic testing at or near the site of patient care) testing for HPV. Researchers are interested in evaluating both tests to determine the best strategy for HPV testing of women who live in rural or underserved areas that have a high prevalence of cervical cancer diagnoses.

Objectives:

* To evaluate the clinical performance of the HPV E6 Test and careHPV in detecting cervical cancer and precancerous lesions.
* To evaluate the best low-cost test or combination of tests for women who have been referred for cervical cancer screening or treatment.
* To compare the clinical performance of self-collected specimens versus clinician-collected specimens in detecting cervical cancer and precancerous lesions.

Eligibility:

- Women between 25 and 65 years of age who live in rural China.

Design:

* This study involves an initial testing visit and a 1-year followup visit for a high-risk subgroup.
* Participants will have the HPV E6 test, careHPV, and a visual inspection test for cervical cancer. For comparison, participants will also have the standard HPV test approved by the U.S. Food and Drug Administration.
* Participants who test positive for HPV on any of the above tests will also have colposcopy to collect samples of cervical tissue for further study.
* A random sample of women who test negative for HPV will also have colposcopy. Participants may also have biopsies if there is visual evidence of cervical abnormalities.
* At the 1-year followup visit, participants in the high-risk subgroup will have the same tests as in the previous visit..

DETAILED DESCRIPTION:
Low-cost, molecular human papillomavirus (HPV) testing may offer a more robust alternative to Pap smears and visual inspection with acetic acid (VIA) for cervical cancer screening of underserved women. Two low-cost molecular tests for human papillomavirus (HPV) have been developed: 1) AVantage HPV E6 Test (Arbor Vita Corporation, Sunnyvale, CA, USA) ( HPV E6 Test ) detects E6 oncoproteins from HPV16, 18, and 45 and 2) careHPV (Qiagen, Gaithersburg, MD, USA) detects the DNA for a pool of 14 carcinogenic HPV genotypes. The HPV E6 Test will be ready for the first clinical evaluations in 2010. The HPV E6 Test works like an ELISA in strip format such that it takes less than two hours to run and may provide point-of-care (diagnostic testing at or near the site of patient care) testing. careHPV, a batch HPV DNA test that takes 2.5 hours to perform, has already been developed and is currently being used in demonstration projects. The results to date for careHPV are promising. As our primary objective, we wish to evaluate both tests, and to evaluate the best low-cost triage strategies for careHPV-positive results in areas of high prevalence of carcinogenic HPV DNA. A study of 7,500 women, ages 25-65 years, identified from an age- and region-stratified sample of women living in rural China will be conducted. All women will be screened at enrollment, and a high-risk subgroup at the one-year follow-up, by the following tests: HPV E6 Test, careHPV, and visual inspection with acetic acid (VIA). Women will also be screened at enrollment, and a high-risk subgroup at the one-year follow-up, using the digene HC2 HPV DNA Test TM ( HC2 ) (formerly known as Hybrid Capture 2)(Qiagen), the first U.S. Food and Drug Administration-approved HPV test and the gold standard for clinical HPV testing. At both time points, all screen-positive women will be evaluated by colposcopy using a rigorous diagnostic protocol. A random sample of screen negatives will undergo colposcopy but will only undergo biopsies if there is visual evidence of cervical epithelial abnormalities. careHPV-positive specimens will be tested for most carcinogenic HPV genotypes, HPV16, HPV18, and HPV45 using careHPV16/18/45. This triage test utilizes the same test platform as careHPV but screens only for those 3 carcinogenic HPV genotypes. The primary goals are 1) to evaluate the clinical performance of careHPV, the HPV E6 Test, and VIA for detection of cervical precancer and cancer and 2) to determine the positive predictive values of VIA, the HPV E6 Test, and HPV16/18/45 detection by careHPV16/18/45 for cervical precancer and cancer among careHPV-positive women.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. have not been previously diagnosed with cervical cancer
  2. have a cervix
  3. are not pregnant
  4. are physically able to undergo routine cervical cancer screening 5) are able to provide informed consent
* We will not exclude women if they have had previous cervical cancer screening because we assume that even if a few women have been screened for cervical cancer, the quality of cytology screening was very poor.

EXCLUSION CRITERIA:

1) are not married AND report never having had sexual intercourse 2) have had a total hysterectomy

3) have a history of cervical cancer

4) are physically or mentally unable to undergo routine cervical cancer screening or unable to provide informed consent.

5) are pregnant or have been pregnant in the last month

-Women who are currently menstruating at the time of enrollment will be deferred from participating, and will become eligible to participate 7-14 days after menstruation has ended. The menstruating women will be advised to return for the screening 7 to 14 days after their menstrual period has concluded.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7500 (Estimated)
Dates: Start 2010-10-11; Study Completion 2010-12-20

CONTACTS AND LOCATIONS:
Locations (2):
- PATH, Seattle, Washington, United States
- CICAMS, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Doorbar J. Molecular biology of human papillomavirus infection and cervical cancer. Clin Sci (Lond). 2006 May;110(5):525-41. doi: 10.1042/CS20050369. PMID 16597322
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Munoz N, Castellsague X, Berrington de Gonzalez A, Gissmann L. Chapter 1: HPV in the etiology of human cancer. Vaccine. 2006 Aug 31;24 Suppl 3:S3/1-10. doi: 10.1016/j.vaccine.2006.05.115. Epub 2006 Jun 23. PMID 16949995
- [Derived] Zhao FH, Jeronimo J, Qiao YL, Schweizer J, Chen W, Valdez M, Lu P, Zhang X, Kang LN, Bansil P, Paul P, Mahoney C, Berard-Bergery M, Bai P, Peck R, Li J, Chen F, Stoler MH, Castle PE. An evaluation of novel, lower-cost molecular screening tests for human papillomavirus in rural China. Cancer Prev Res (Phila). 2013 Sep;6(9):938-48. doi: 10.1158/1940-6207.CAPR-13-0091. Epub 2013 Jul 22. PMID 23878179